CLINICAL TRIAL: NCT03313245
Title: Diet Quality and Cognitive Control Function in Early Childhood: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, Naiman Khan, Assistant Professor, University of Illinois at Urbana-Champaign
Other Study IDs: 16484
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Diet Habit; Cognitive Function
MeSH Terms: conditions — Feeding Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention/Observational Study — No Intervention/Observational Study

SUMMARY:
This study aims to study the relationship between diet and cognitive function among 4-5-year-olds.

DETAILED DESCRIPTION:
Children's ability for optimal cognitive function is critical for their long-term capacity to learn and achieve scholastic success. However, there is a gap in the knowledge pertaining to the selection of appropriate cognitive tasks for studying relationships between diet and cognitive control, particularly among young children. Accordingly, this study aims to study the relationship between diet and cognitive function using a standardized neuropsychological assessment and a modified cognitive task battery.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* Child Assent
* 4 and 5 years of age
* Absence of neurological disorders
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Younger than 4 and older than 5 years of age
* Presence of neurological disorders
* Uncorrected vision

Ages: 4 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: 4 and 5-year-olds
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Cognitive and Academic Development | Once at laboratory visit
  Woodcock Johnson IV eCAD

SECONDARY OUTCOMES:
Attention | Once at laboratory visit
  2-stimulus Oddball task
Cognitive Flexibility | Once at laboratory visit
  Hearts and Flowers Task
Diet Quality | 7-day average following first laboratory visit
  Healthy Eating Index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology and Community Health, Urbana, Illinois, United States